CLINICAL TRIAL: NCT03951064
Title: Effect of Esophageal Pressure Measurement to Determine Optimal Positive End-expiratory Pressure Compared to Usual Care in Obese Patients Receiving Mechanical Ventilation
Brief Title: Providing Optimal PEEP During Mechanical Ventilation for Obese Patients Using Esophageal Balloon
Acronym: PROP OPEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Since November 2022, an indefinite pause of study activities caused by a hospital-wide shortage of esophageal balloons has persisted for almost a full year with an indefinite resupply date. Thus, the PI has opted to close to any further enrollment.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-2010
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid; Ventilator-Induced Lung Injury; Respiratory Failure
Keywords: Transpulmonary pressure; Esophageal balloon; Esophageal pressure monitoring; Mechanical ventilation
MeSH Terms: conditions — Obesity, Morbid; Ventilator-Induced Lung Injury; Respiratory Insufficiency | interventions — Serum Bactericidal Test; Airway Extubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the obvious treatment differences between the two groups, blinding of treatment group will be impossible. However, the investigators will have one outcome assessor who will have access only to the data necessary to determine the primary outcome (Ventilator-Free Days at 28-days), and this assessor will be blinded to treatment group using built-in REDCap tools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Optimal PEEP (Experimental): The waveforms of airway pressure (Paw), esophageal pressure (Pes), and transpulmonary pressure (Ptp) will be visualized on the ventilator. Ptp is obtained from Paw - Pes. PEEP will be increased on the ventilator to achieve a Ptp between 0 and +2 cm H2O (Optimal PEEP). Measurements will be obtained daily and adjustments to PEEP will occur daily. PEEP will be reduced below Optimal PEEP in the setting of hemodynamic compromise (requiring increasing vasoactive medications for blood pressure support).
  Interventions: Device: Esophageal balloon; Procedure: Intervention Spontaneous Breathing Trial (SBT) and Extubation; Procedure: Intervention Weaning after Tracheostomy
- Acute Hypoxic Respiratory Distress Syndrome Network (ARDSNet) High PEEP (Active Comparator): PEEP in the control group will be determined by High PEEP ARDSnet PEEP/FiO2 table. Titration of PEEP will occur when clinically indicated by partial pressure of oxygen (PaO2) or oxygen saturation (SpO2), and FiO2. The investigators chose the High PEEP table based on the clinical suspicion that obese patients may require higher PEEP levels on average than non-obese patients to balance the additional pressure of their chest wall. In addition, EPVent2, a study of esophageal balloon PEEP titration in patients with ARDS utilized the High PEEP table. Patients with moderate and severe ARDS benefit from higher levels of PEEP.
  Interventions: Device: Esophageal balloon; Procedure: Control Spontaneous Breathing Trial and Extubation; Procedure: Control Weaning after Tracheostomy

INTERVENTIONS:
Device: Esophageal balloon — All patients in both groups will have an esophageal balloon catheter inserted by a research investigator. The catheter will be inserted into their nare while upright (head of bed >30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Gastric positioning will be confirmed with abdominal compression testing and the catheter then retracted 10 - 20cm into the lower esophagus. Placement will be confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the patient's nasal opening using tape.
Procedure: Intervention Spontaneous Breathing Trial (SBT) and Extubation — Patients in the Intervention group will undergo an SBT regardless of their PEEP level. The PEEP that generates a Ptp of 0 will be considered their optimal PEEP, and this will not be lowered for the SBT. The Intervention Group SBT will consist of a trial of a pressure support of 5 cm H2O and Optimal PEEP.
  Arms: Optimal PEEP
Procedure: Control Spontaneous Breathing Trial and Extubation — Patients in the Control group will undergo an SBT when they reach a PEEP ≤8 cm H2O. This is the current standard of care based on the SBT protocol at UNC Hospitals. SBT and extubation prior to meeting these criteria will be based on primary medical team's discretion and will be recorded for analysis and safety tracking.
  Arms: Acute Hypoxic Respiratory Distress Syndrome Network (ARDSNet) High PEEP
Procedure: Intervention Weaning after Tracheostomy — Based on the use of optimal PEEP in this group, and the experience in the previous study protocol, the investigators will place patients in the Intervention group on Tracheostomy Collar Trial only with a speaking valve. This simulates the normal process of utilizing the upper airway to maintain lung inflation that is performed automatically when a patient does not have an artificial airway.
  Arms: Optimal PEEP
Procedure: Control Weaning after Tracheostomy — The control group will be placed on Tracheostomy Collar Trial with no requirement for speaking valve. They may utilize a speaking valve if tolerated and desired, but there is no requirement as there is in the Intervention group.
  Arms: Acute Hypoxic Respiratory Distress Syndrome Network (ARDSNet) High PEEP

SUMMARY:
This is a research study to determine if identifying an optimal level of positive end-expiratory pressure (PEEP) targeted specifically to individualized patient characteristics will shorten the time on the ventilator.

Participants will have catheter placed through the nose into the esophagus to measure the pressure inside the chest. This catheter will remain until the patient is freed from the ventilator. Participants will be randomized to usual care or to have the level of PEEP determined by the esophageal balloon pressure readings. The total time spent on the ventilator will be recorded.

DETAILED DESCRIPTION:
Study Design:

Randomized-controlled clinical trial. Patients will be enrolled within 4 days of mechanical ventilation and randomized 1:1 to titration of PEEP based on esophageal balloon pressures or based on the "High PEEP" ARDSnet PEEP/fraction of inspired oxygen (FiO2) table. All patients will have esophageal balloons placed with baseline measurement of Ptp. Patients randomized to the intervention arm will then undergo titration of PEEP based on Ptp measurements to achieve "Optimal PEEP," defined as end expiratory Ptp of 0 to +2 cm water (H2O).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 40
* Acute respiratory failure requiring mechanical ventilation

Exclusion Criteria:

* Refusal to give consent by the subject or their legally authorized representative
* Abdominal compartment syndrome
* Chest tube for pneumothorax
* Having been on a ventilator for >4 days
* Suspicion of or known intracranial hypertension
* Anticipated extubation within 24 hours
* Chronic ventilator dependence
* Condition that precludes placement of an esophageal balloon (esophageal or nasopharyngeal pathology preventing insertion of the esophageal balloon catheter, severe thrombocytopenia or coagulopathy)
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Carson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset will be available to investigators 9-36 months following publication of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: Data can be obtained upon application to primary investigators. Investigators who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Obi ON, Mazer M, Bangley C, Kassabo Z, Saadah K, Trainor W, Stephens K, Rice PL, Shaw R. Obesity and Weaning from Mechanical Ventilation-An Exploratory Study. Clin Med Insights Circ Respir Pulm Med. 2018 Sep 18;12:1179548418801004. doi: 10.1177/1179548418801004. eCollection 2018. PMID 30245572
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimal Post End Expiratory Pressure (PEEP): Obese adult participants presenting to the ICU with acute respiratory failure requiring mechanical ventilation were enrolled. Mechanical ventilation settings were monitored daily and Post End Expiratory Pressure (PEEP) setting adjusted based on the balloon measurements.
  Esophageal balloon: Participants will have an esophageal balloon catheter inserted by a research investigator. The catheter will be inserted into the nare while upright (head of bed >30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Placement confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the nasal opening using tape.
  Intervention Spontaneous Breathing Trial (SBT) and Extubation: Participants undergo an SBT regardless of PEEP level. The PEEP that generates a Ptp of 0 was considered the optimal PEEP, and this will not be lowered for the SBT. The Intervention Group SBT will consist of a trial of a pressure support of 5 cm water (H2O) and Optimal PEEP.
  Intervention Weaning after Tracheostomy: Based on the use of optimal PEEP in this group and the experience in the previous study protocol, the investigators will place participants in the Intervention group on Tracheostomy Collar Trial only with a speaking valve.
- ARDSNet High PEEP: Obese adult participants presenting to the ICU with acute respiratory failure requiring mechanical ventilation were enrolled. PEEP in the control group will be determined by High PEEP ARDSnet PEEP/FiO2 table. Titration of PEEP will occur when clinically indicated by partial pressure of oxygen (PaO2) or oxygen saturation (SpO2), and fraction of inspired oxygen (FiO2)
  Esophageal balloon: Participants will have an esophageal balloon catheter inserted by a research investigator. The catheter will be inserted into the nare while upright (head of bed >30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Placement confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the nasal opening using tape.
  Control Spontaneous Breathing Trial and Extubation: Participants in the Control group will undergo an SBT when they reach a PEEP ≤8 cm H2O. SBT and extubation prior to meeting these criteria will be based on primary medical team's discretion and will be recorded for analysis and safety tracking.
  Control Weaning after Tracheostomy: The control group will be placed on Tracheostomy Collar Trial with no requirement for speaking valve. They may utilize a speaking valve if tolerated and desired, but there is no requirement as there is in the Intervention group.
Period: Overall Study
Arm/Group | Optimal Post End Expiratory Pressure (PEEP) | ARDSNet High PEEP
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Optimal PEEP: Obese adult participants presenting to the ICU with acute respiratory failure requiring mechanical ventilation were enrolled. Mechanical ventilation settings were monitored daily and PEEP setting adjusted based on the balloon measurements.
  Esophageal balloon: Participants will have an esophageal balloon catheter inserted by a research investigator. The catheter will be inserted into the nare while upright (head of bed >30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Placement confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the nasal opening using tape.
  Intervention Spontaneous Breathing Trial (SBT) and Extubation: Participants undergo an SBT regardless of PEEP level. The PEEP that generates a Ptp of 0 was considered the optimal PEEP, and this will not be lowered for the SBT. The Intervention Group SBT will consist of a trial of a pressure support of 5 cm H2O and Optimal PEEP.
  Intervention Weaning after Tracheostomy: Based on the use of optimal PEEP in this group, and the experience in the previous study protocol, the investigators will place participants in the Intervention group on Tracheostomy Collar Trial only with a speaking valve. This simulates the normal process of utilizing the upper airway to maintain lung inflation that is performed automatically when a participant does not have an artificial airway.
- ARDSNet High PEEP: Obese adult participants presenting to the ICU with acute respiratory failure requiring mechanical ventilation were enrolled. PEEP in the control group will be determined by High PEEP ARDSnet PEEP/FiO2 table. Titration of PEEP will occur when clinically indicated by partial pressure of oxygen (PaO2) or oxygen saturation (SpO2), and FiO2
  Esophageal balloon: Participants will have an esophageal balloon catheter inserted by a research investigator. The catheter will be inserted into the nare while upright (head of bed >30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Placement confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the nasal opening using tape.
  Control Spontaneous Breathing Trial and Extubation: Participants in the Control group will undergo an SBT when they reach a PEEP ≤8 cm H2O. SBT and extubation prior to meeting these criteria will be based on primary medical team's discretion and will be recorded for analysis and safety tracking.
  Control Weaning after Tracheostomy: The control group will be placed on Tracheostomy Collar Trial with no requirement for speaking valve. They may utilize a speaking valve if tolerated and desired, but there is no requirement as there is in the Intervention group.
- Total: Total of all reporting groups
Arm/Group | Optimal PEEP | ARDSNet High PEEP | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventilator-Free Days (VFD) by Day 28
Description: The number of days a patient is alive and free from the ventilator up to day 28.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
Days | 2.33 (5.86) | 6.67 (13.32)

2. Secondary Outcome: Number of Participants Reintubated
Description: Intubated within 72 hours of extubation
Time Frame: 72 hours after extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
Participants | 2 | 1

3. Secondary Outcome: ICU Length of Stay
Description: Number of days spent in the ICU
Time Frame: maximum duration of ICU stay, up to 46 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
Days | 37.33 (7.77) | 24.00 (18.33)

4. Secondary Outcome: Hospital Length of Stay
Description: Number of days spent in the Hospital
Time Frame: maximum duration of hospital stay, up to 83 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
Days | 62.67 (18.45) | 33.67 (29.02)

5. Secondary Outcome: Number of Patients Receiving a Tracheostomy
Description: Whether the patient required a tracheostomy to be liberated from the ventilator
Time Frame: during mechanical ventilation, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

6. Secondary Outcome: Number of Patients Extubated Early
Description: Extubation prior to meeting established criteria (Control group only). Participants in the Control group will undergo an SBT when they reach a PEEP ≤8 cm H2O. This is the current standard of care based on the SBT protocol at UNC Hospitals. SBT and extubation prior to meeting these criteria will be based on primary medical team's discretion and will be recorded for analysis and safety tracking.
Time Frame: 28 days
Population: This measure only applies to the Control group. These data were not collected for the Optimal PEEP arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 0 | 3
Participants |  | 2

7. Secondary Outcome: Highest Richmond Agitation and Sedation Scale
Description: Measures the mental and physical state of a sedated patient. Range from -5 to +4. A score of 0 indicates a calm arousable patient and is the ideal score. A score of +4 indicates a very combative participant and a score of -5 indicates an unarousable participant. This outcome captures the highest score measured throughout mechanical ventilation with scores on the extreme ends of the range reflecting a worse outcome.
Time Frame: during mechanical ventilation, up to 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
score on a scale | 2.33 (0.58) | 2.00 (0.00)

8. Secondary Outcome: Lowest Richmond Agitation and Sedation Scale
Description: Measures the mental and physical state of a sedated patient. Range from -5 to +4. A score of 0 indicates a calm arousable patient and is the ideal score. A score of +4 indicates a very combative participant and a score of -5 indicates an unarousable participant. This outcome captures the lowest score measured throughout mechanical ventilation with scores on the extreme ends of the range reflecting a worse outcome.
Time Frame: during mechanical ventilation, up to 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Optimal PEEP | ARDSNet High PEEP
Number analyzed (Participants) | 3 | 3
score on a scale | -4.67 (0.58) | -4.67 (0.58)

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent through 28 days of mechanical ventilation or successful extubation (whichever occurred first).
Arm/Group | Optimal PEEP | ARDSNet High PEEP
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal PEEP (N=3) | ARDSNet High PEEP (N=3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal PEEP (N=3) | ARDSNet High PEEP (N=3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Diagnosed during study
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated creatinine kinase (Renal and urinary disorders) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT03951064/Prot_SAP_000.pdf